CLINICAL TRIAL: NCT03577743
Title: Phase 2 Study to Evaluate the Effect of Bevacizumab in Metastatic Triple Negative Breast Cancer
Brief Title: Effect of Bevacizumab in Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebat-Allah Mahmoud Bakri Ahmed, assisstant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTN
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Triple Negative Breast Cancer; Safety Issues; Efficacy
Keywords: antiangiogenesis; taxanes and carboplatin; metastatic TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): bevacizumab and chemotherapy given every 21 day untill disease progression or unacceptable toxicity
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — -bevacizumab 15m.g/ kg + carboplatin 450m.g + paclitaxel 175m.g/m2 D1 /21 Day until disease progression or un acceptable toxicity .
  Other Names: avastin

SUMMARY:
Evaluating efficacy and safety of bevacizumab when combined with chemotherapy (carboplatin and Paclitaxel ) in treatment of patient with metastatic triple negative breast cancer

DETAILED DESCRIPTION:
Breast cancer is the most common non cutaneous cancer in U.S. women, with an estimated 63,960 cases of in situ disease and 266,120 cases of invasive disease in 2018. (American Cancer Society: Cancer Facts and Figures 2018). On the basis of ER, PR, and HER2/neu results, breast cancer is classified as one of the following types:

Hormone receptor positive , HER2/neu positive and Triple negative (ER, PR, and HER2/neu negative).

ER, PR, and HER2 status are important in determining prognosis and in predicting response to endocrine and HER2-directed therapy.(Harris JR, Morrow M, Lippman ME, et al . 1996) Metatstaic Triple-negative breast cancer (TNBC) is a diagnosis of exclusion, defined by the lack of expression of estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER2) .

TNBC tends to occur in younger, often premenopausal patients, African Americans, and in association with hereditary syndromes, most commonly germline BRCA1 mutations. It constitutes up to 15% of all breast cancers but accounts for > 25% of breast cancer-related deaths as it has an inherent predisposition for rapid dissemination and visceral metastases with limited improvements in overall survival and inferior clinical outcomes . It is characterized by higher incidence of brain metastases and rapid progression from the onset of metastasis to death. Having aggressive biology more than other breast types due to high risk of early relapse between the first and third years after diagnosis , metastases are rarely preceded by local recurrence and most deaths occur in the first 5 years ( Livasy CA et al . 2006 ) Due to the palliative intent of treatment as in MBC and Optimal chemotherapy regimens have yet to be established in treatment of metastatic TNBC; however, there have been advances in the systemic treatment of triple-negative breast cancer in the neoadjuvant, adjuvant, and metastatic settings. ( J.M. Lebert , R. Lester , E. Powell et el current oncology journal 2018 ) it is critical that an individualized approach is taken that incorporates patient, disease, and treatment-related factors, including an individual oncologist treatment preference.(Geels P, et al 2000 ).

There have been several head-to-head chemotherapy trials performed within the metastatic setting, and much of what is applied in clinical practice is extrapolated from chemotherapy trials in the adjuvant setting, with taxanes and anthracyclines incorporated early on in the patient's treatment course.

Angiogenesis is essential for the development of malignancies and plays a central role in the early stages of growth, invasion, and metastatic spread of breast cancer (BC), thus representing a reasonable therapeutic target. This evidence is a solid biological rationale for the use of therapeutic agents able to interfere with the VEGF (vaso endothelial growth factor ) function.

Breast cancer is the most common non cutaneous cancer in U.S. women, with an estimated 63,960 cases of in situ disease and 266,120 cases of invasive disease in 2018. (American Cancer Society: Cancer Facts and Figures 2018). On the basis of ER, PR, and HER2/neu results, breast cancer is classified as one of the following types:

Hormone receptor positive , HER2/neu positive and Triple negative (ER, PR, and HER2/neu negative).

ER, PR, and HER2 status are important in determining prognosis and in predicting response to endocrine and HER2-directed therapy.(Harris JR, Morrow M, Lippman ME, et al . 1996) Metatstaic Triple-negative breast cancer (TNBC) is a diagnosis of exclusion, defined by the lack of expression of estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER2) .

TNBC tends to occur in younger, often premenopausal patients, African Americans, and in association with hereditary syndromes, most commonly germline BRCA1 mutations. It constitutes up to 15% of all breast cancers but accounts for > 25% of breast cancer-related deaths as it has an inherent predisposition for rapid dissemination and visceral metastases with limited improvements in overall survival and inferior clinical outcomes . It is characterized by higher incidence of brain metastases and rapid progression from the onset of metastasis to death. Having aggressive biology more than other breast types due to high risk of early relapse between the first and third years after diagnosis , metastases are rarely preceded by local recurrence and most deaths occur in the first 5 years ( Livasy CA et al . 2006 ) Due to the palliative intent of treatment as in MBC and Optimal chemotherapy regimens have yet to be established in treatment of metastatic TNBC; however, there have been advances in the systemic treatment of triple-negative breast cancer in the neoadjuvant, adjuvant, and metastatic settings. ( J.M. Lebert , R. Lester , E. Powell et el current oncology journal 2018 ) it is critical that an individualized approach is taken that incorporates patient, disease, and treatment-related factors, including an individual oncologist treatment preference.(Geels P, et al 2000 ).

There have been several head-to-head chemotherapy trials performed within the metastatic setting, and much of what is applied in clinical practice is extrapolated from chemotherapy trials in the adjuvant setting, with taxanes and anthracyclines incorporated early on in the patient's treatment course.

Angiogenesis is essential for the development of malignancies and plays a central role in the early stages of growth, invasion, and metastatic spread of breast cancer (BC), thus representing a reasonable therapeutic target. This evidence is a solid biological rationale for the use of therapeutic agents able to interfere with the VEGF (vaso endothelial growth factor ) function.

The recombinant monoclonal antibody bevacizumab is currently the most widely used and developed antiangiogenic drug in the treatment of breast cancer(BC) , able to recognize all the isoforms of VEGFA, preventing its binding to the cellular receptor, and inhibiting the angiogenic and proliferative signal. In vivo studies showed that bevacizumab inhibits both proliferation and migration of endothelial cells induced by VEGFA; besides in some models of human BC, the treatment with bevacizumab was associated to a reduction in microvascular density ( Zhang W et al. 2002. ) . The humanized, anti-VEGF monoclonal antibody bevacizumab has been shown to increase progression-free survival (PFS) and/ or overall survival (OS) in metastatic breast cancer (MBC), response rate RR . ( Brufsky A, et al 2012) ( Vrdoljak E1, et al 2016 ).

In the Phase 3 RIBBON-2 study, previously treated patients with metastatic breast cancer were randomized to Avastin with chemotherapy (n=112 had triple-negative breast cancer) or chemotherapy with placebo (n=47 had triple-negative breast cancer). In an exploratory subgroup analysis of the patients with triple-negative breast cancer, median progression-free survival was 6 months vs 2.7 months (hazard ratio=0.49; p=0.0006), median overall survival was 17.8 months vs 13.5 months (hazard ratio=0.85; 95% CI, 0.58-1.26), and objective response rate was 41% vs 18% (p=0.0078). (Brufsky AM, Hurvitz S, Perez E, et al. 2012 ) In the RIBBON-1 study, chemotherapy with or without Avastin was evaluated in 1,237 patients as first-line treatment for metastatic breast cancer, 21.3% of whom had triplenegative breast cancer. In prespecified subgroup analyses, triple-negative patients demonstrated a hazard ratio for progression-free survival of 0.72 (95% CI, 0.49-1.06) and had a median progression-free survival of 6.1 vs. 4.2 months in the Avastin with capecitabine arm vs the capecitabine alone arm. In the Avastin with taxane/anthracycline cohort vs taxane/anthracycline alone cohort, triple-negative patients had a hazard ratio for progressionfree survival of 0.78 (95% CI, 0.53-1.15) with a median progression-free survival of 6.5 vs 6.2 months, respectively. (Robert NJ, Diéras V, Glaspy J, et al. RIBBON-1 ,2011) A subgroup analysis of the TURANDOT study compared first-line Avastin and paclitaxel (Arm A) with Avastin and capecitabine (Arm B) in human epidermal growth factor receptor 2-negative patients with triple-negative metastatic breast cancer (n=124). In the triplenegative breast cancer subgroup, the median overall survival was 24.4 months in Arm A and 17.7 months in Arm B (unstratified hazard ratio=1.35; 95% CI, 0.9-2.02). (Zielinski C, Lang I, Inbar M, et al. 2016) Taxanes as part of chemotherapy have been studied as having an inhibitory action on the proliferation of endothelial progenitor cells, with an antiangiogenic effect at lower doses than those needed to inhibit the proliferation of cancer cells. The resulting hypoxia induces cancer cells to a kind of "reaction" through the autocrine production of proangiogenic agents , several evidences of their benefits on clinical outcomes, such as OS, time to progression (TTP), and over all response rate ( ORR.) ( Tran J. et al. 2002.) ( Ghersi D, et al. 2015 ) . Even if conventional taxanes demonstrated to be more active in endocrine receptor-negative tumors and are indicated in the first-line treatment of TNBC . ( Isakoff SJ Cancer J. 2010 ) Because of the sensitivity of TNBC to platinum compounds and the synergistic effect of bevacizumab with paclitaxel we investigated the efficacy and toxicity of weekly paclitaxel and carboplatin in combination with bevacizumab as first-line treatment in metastatic TNBC.

phase II study followed the Simon's 2-stage optimal design. Paclitaxel (90 mg/m2) and carboplatin (2 area under the curve) were administered on days 1, 8, and 15 every 4 weeks, preceded by bevacizumab 10 mg/kg on days 1 and 15. The primary end point was the objective response rate (ORR). A total of 46 patients were enrolled. Seven (15.2%) complete and 23 (50%) partial responses were observed for an ORR of 65.2% (95% confidence interval, 52.9%-80.4%). The median progression-free survival was 10.3 months, the median overall survival 25.7 months, and the median duration of response 18.2 months. Neutropenia Grade III and IV was experienced by 13 (28.3%) and 6 (13.04%) patients, respectively. One patient developed an uneventful Grade IV thrombocytopenia. There was 1 toxic death due to febrile neutropenia. Other Grade III toxicities included anemia (n = 2), neurotoxicity (n = 2), thrombocytopenia (n = 1), and diarrhea (n = 1). No serious bevacizumab-related toxicities were observed.( Saloustros E, Nikolaou M, Kalbakis etal 2017)

ELIGIBILITY:
Inclusion Criteria:

1. Female patient firstly diagnosed with metastatic TNBC or after adjuvant treatment OF TNBC by immune histochemistry and biopsy
2. Age >18 Y
3. Performance status (PS ) 0-2
4. Did not have any bleeding disorders.
5. Receive only one line of chemotherapy in adjuvant ttt

Exclusion Criteria:

1. Male patient
2. PS >2
3. Uncontrolled HPTN
4. Have history of bleeding disorders
5. Receive > one line of chemotherapy
6. Have other type of malignancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
- progression free survival | after six month from last enrollment
  the length of time during and after the treatment that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
- Response rate (R.R) : | after 1 year from enrollment
  length of time from the date of diagnosis to the time of death or lost follow up.
- Over all survival. | after 3 years
  the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: assuit university, Study Director — Assiut University
Locations (1):
- Clinical Oncology Departement Assuit University Hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brufsky A, Valero V, Tiangco B, Dakhil S, Brize A, Rugo HS, Rivera R, Duenne A, Bousfoul N, Yardley DA. Second-line bevacizumab-containing therapy in patients with triple-negative breast cancer: subgroup analysis of the RIBBON-2 trial. Breast Cancer Res Treat. 2012 Jun;133(3):1067-75. doi: 10.1007/s10549-012-2008-6. Epub 2012 Mar 14. PMID 22415477
- [Result] Zielinski C, Lang I, Inbar M, Kahan Z, Greil R, Beslija S, Stemmer SM, Zvirbule Z, Steger GG, Melichar B, Pienkowski T, Sirbu D, Petruzelka L, Eniu A, Nisenbaum B, Dank M, Anghel R, Messinger D, Brodowicz T; TURANDOT investigators. Bevacizumab plus paclitaxel versus bevacizumab plus capecitabine as first-line treatment for HER2-negative metastatic breast cancer (TURANDOT): primary endpoint results of a randomised, open-label, non-inferiority, phase 3 trial. Lancet Oncol. 2016 Sep;17(9):1230-9. doi: 10.1016/S1470-2045(16)30154-1. Epub 2016 Aug 5. PMID 27501767
- [Result] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Derived] Mohamed RF, Bakri HM, Abdelfattah ON, Eid S. Does bevacizumab carry a hope for metastatic triple-negative breast cancer in the era of immunotherapy? Anticancer Drugs. 2022 Jan 1;33(1):e604-e609. doi: 10.1097/CAD.0000000000001192. PMID 34407054
- Available data/document: Study Protocol: BMTN — http://clinicaltrials.gov/NCT03577743 — Phase 2 study to evaluate the effect of bevacizumab in metastatic triple negative breast cancer patients